CLINICAL TRIAL: NCT05922852
Title: the Effect of Novel Antidiabetic Drug Combined With Angiotensin Receptor/Neprilysin Inhibitor Over Monotherapy on Urinary Protein in Patients With Type 2 Diabetes
Brief Title: Effect of Novel Antidiabetic Drug Combined With Angiotensin Receptor/Neprilysin Inhibitor on Urinary Protein
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023228
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; Antidiabetic Drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SGLT2i+ARNI: patients in this group received SGLT2i combined with ARNI medication。
- SGLT2i only: patients in this group received SGLT2i medication only。
- ARNI only: patients in this group received ARNI medication only。
- control: patients in this group received neither SGLT2i nor ARNI。

SUMMARY:
The purpose of this study is to determine whether the combination of SGLT2i and ARNI in type 2 diabetic patients with combined albuminuria could reduce urinary protein more significantly than single agent.

DETAILED DESCRIPTION:
This project is a single-center retrospective cohort study to obtain the biochemical index levels of urinary albumin creatinine ratio, urinary protein creatinine ratio, blood renal function, blood lipids, and blood glucose at the immediate, 3rd, 6th, and 12th month of cohort inclusion in each group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Clinical diagnosis of type 2 diabetes mellitus
* Immediate urine albumin creatinine ratio greater than 30mg/g
* Signed informed consent and available for follow-up

Exclusion Criteria:

* severe renal insufficiency, i.e. eGFR ≤ 30ml/min/1.75m2
* clinical diagnosis of various acute and chronic urinary tract infections
* combined with various serious infectious diseases
* combined with acute complications of diabetes mellitus
* end-stage malignancy
* pregnancy and lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
urinary protein changes | 2023.03-2024.03
  to determine whether the combination of SGLT2i and ARNI in type 2 diabetic patients with combined albuminuria could reduce urinary protein more significantly than single agent.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing 100191, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Xu L, Chen B, Zhang H, Zhu D. Combined effects of sodium-glucose cotransporter 2 inhibitor and angiotensin receptor-neprilysin inhibitor on renal function in cardiovascular disease patients with type 2 diabetes mellitus: a retrospective cohort study. Front Endocrinol (Lausanne). 2024 Jan 11;14:1326611. doi: 10.3389/fendo.2023.1326611. eCollection 2023. PMID 38274236